CLINICAL TRIAL: NCT00820157
Title: A Prospective Randomized Trial Comparing Cytoreductive Surgery Followed by Transcatheter Arterial Chemoembolization (TACE) Versus TACE Alone for Multinodular Hepatocellular Carcinoma (MNHCC)
Brief Title: Cytoreductive Surgery and Transarterial Chemoembolization (TACE) Versus TACE for Hepatocellular Carcinoma
Acronym: TACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-021
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma, Hepatocellular; Chemoembolization, Therapeutic; Cytoreductive
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cytoreductive Surgery (Active Comparator): Cytoreductive Surgery followed by TACE
  Interventions: Procedure: Cytoreductive Surgery
- TACE (Experimental): TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: Cytoreductive Surgery — Cytoreductive Surgery followed by TACE for MNHCC
  Other Names: Cytoreductive group
  Arms: Cytoreductive Surgery
Procedure: TACE — TACE alone or TACE followed by downstage resection for MNHCC
  Other Names: TACE group
  Arms: TACE

SUMMARY:
The aim of this study is to compare the surgical outcomes of cytoreductive surgery followed by Transarterial Chemoembolization (TACE) with TACE alone in patients with MNHCC so as to establish a treatment standard for MNHCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the world's most common malignancies, especially in East-Asian countries. Hepatic resection has been accepted as the only means of cure for patients with HCC. The results of hepatic resection for early-stage HCC are favorable.Nevertheless, the role of surgical resection for multinodular HCC (MNHCC) is less well-defined.The presence of multiple tumors has been shown to be one of the most significant independent factors to influence cumulative survival rates in HCC after hepatic resection.Using the BCLC criteria,liver transplantation provides an alternative curative treatment option for MNHCC with size ≤ 5 cm in diameter and tumor number <3，but MNHCC beyond these criteria usually receive palliative therapy.

For MNHCC which not suitable for curative treatment, non-surgical and surgical interventions are available for palliative care.Cytoreductive surgery has the potential to increase the quality and quantity of survival in patients with advanced HCC. Cytoreductive surgery is carried out with partial hepatectomy,cryosurgery,microwave coagulation therapy(MCT),or absolute alcohol injection.It has been shown to prolong survival and provide good symptomatic relief in patients with good surgical risks in non-randomized studies.Cytoreductive surgery aims at removal or destruction of all macroscopic tumours, allowing microscopic foci to persist while preserving as much of the functional liver tissue as possible. The development of effective local ablative therapy (LAT), such as radiofrequency ablation (RFA) therapy, facilitates reduction of the tumour burden even further during the operation.Cytoreductive surgery can also be followed by other non-surgical treatments,such as regional therapy or systemic therapy, to deal with the residual disease or micrometastases.

The aim of this study is to compare the surgical outcomes of cytoreductive surgery followed by TACE with TACE alone in patients with MNHCC so as to establish a treatment standard for MNHCC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* at least 2 radiologic imaging showing characteristic features of HCC or one radiologic imaging associated with AFP >400 or cytologic/histologic evidence.
* tumor number >3 and <=5,maximum diameter >5cm and <=15cm;without evidence of radiologically definable vascular invasion or extrahepatic metastasis.
* Criteria of liver function: Child A-B level, serum bilirubin ≤ 1.5 times the upper limit of normal value,alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
* No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal.
* Hb ≥90g/L,WBC ≥3.000 cells/mm³,platelets ≥80.000 cells/mm³
* Patients who can understand this trial and have signed information consent

Exclusion Criteria:

* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer.
* Patients with other diseases which may affect the treatment mentioned.
* Patients with a medical history of other malignant tumors.
* Subjects participating in other clinical trials.
* Extrahepatic metastasis, portal vein or other major vascular involvement.
* liver function:Child C.
* no pathological evidence of HCC.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the overall survival rate of each group | 3 years

SECONDARY OUTCOMES:
the disease-free survival rate of each group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Zhou, M.D., Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China